CLINICAL TRIAL: NCT05867056
Title: An Open-label Study Evaluating the Safety, Antiviral Activity, and Pharmacokinetics of IMC-I109V in HLA-A*02:01 Positive Participants With Chronic HBV Infection Who Are Non-Cirrhotic, Hepatitis B e Antigen-negative, and Virally Suppressed
Brief Title: Study of IMC-I109V in Non-cirrhotic HBeAg-negative Chronic HBV Infection
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Enrollment into the phase 2 portion was never initiated.
Sponsor: Immunocore Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMC-I109V-101; 2019-004212-64 (EudraCT Number)
Record Dates: First submitted 2023-04-12; First posted 2023-05-19 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Hepatitis B, Chronic
Keywords: HBeAg negative; HLA-A*02;01 Positive; T Cell Receptor (TCR)
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — mycophenolic adenine dinucleotide

STUDY DESIGN:
Intervention Model Description: Participants will receive a single dose of IMC-I109V-101 in Part 1 (SAD) and 24 weekly doses in Part 2 (MAD). Participants in Part 3 will receive weekly doses of IMC-I109V until disease progression, unacceptable toxicity, or other reason for treatment discontinuation occurs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Single Ascending Dose (SAD) (Experimental): SAD will be approximately 10 weeks for each participant, comprising a maximum 42-day screening period, a 1-day treatment period involving a single administration of IMC-I109V and a 28-day follow-up period, for a total of 8 visits. Visits will take place on Day -1 and Days 1, 2, 3, 8, 15, 22, and 29. Follow-up may be extended in participants who achieve a decrease in HBsAg of > 0.5 log10 IU/mL at Day 29.
  Interventions: Drug: IMC-I109V Single Ascending Dose
- Part 2: Multiple Ascending Doses (MAD) (Experimental): MAD will be approximately 54 weeks for each participant, comprising a maximum 42-day screening period, a 24-week treatment period involving weekly administration of IMC-I109V, and a 24-week follow-up period, with a total of 29 visits. Visits will take place on Day -1 and Days 1, 3 and 8, Weeks 3 (Day 15) through 24, Weeks 28, 36, 48 and 49. Participants who have achieved HBsAg <100 IU/mL at end of Week 24 may be considered for further study treatments of up to Week 48 and follow-up visits every 12 weeks to Week 72. Treatment will be discontinued at Week 16 in participants who have not shown evidence of a response to IMC-I109V, in order to minimize unnecessary drug exposure in participants who are unlikely to achieve reductions in viral biomarkers with further doses.
  Interventions: Drug: IMC-I109V Multiple Ascending Doses
- Part 3: HBV HCC Module MAD (Experimental): Enrollment into Part 3 may begin at the discretion of the Sponsor and will involve a maximum 42-day screening period, a treatment period comprising weekly administration of the target dose until the criteria for treatment discontinuation are met. Visits will take place on Day 1-2 and Day 8, Week 3 (Day 15), with this cycle being repeated until treatment stops, then 30 and 90 days post-last dose, then every 3 months after last dose, after which there will be a safety follow-up period of 30 days.
  Interventions: Drug: HBV HCC Module MAD

INTERVENTIONS:
Drug: IMC-I109V Single Ascending Dose — Single dose administration of IMC-I109V
  Other Names: SAD
  Arms: Part 1: Single Ascending Dose (SAD)
Drug: IMC-I109V Multiple Ascending Doses — Multidose administration of IMC-I109V
  Other Names: MAD
  Arms: Part 2: Multiple Ascending Doses (MAD)
Drug: HBV HCC Module MAD — Multidose administration of IMC-I109V
  Arms: Part 3: HBV HCC Module MAD

SUMMARY:
IMC-I109V is an immune-mobilizing monoclonal T cell receptor (TCR) against viruses (ImmTAV®), a new class of bispecific protein therapeutics designed for the treatment of chronic hepatitis B virus (HBV) infection (CHB). This is the first in-human study of IMC-I109V in persons with CHB.

DETAILED DESCRIPTION:
IMC-I109V-101 is a first-in-human (FIH) study designed to assess the safety, tolerability, and pharmacokinetic (PK) profile of IMC-I109V in single and multiple dose regimens and to provide a preliminary assessment of antiviral activity, when administered to virally suppressed hepatitis B e-antigen (HBeAg)-negative participants receiving long-term NA therapy. The aim of this study is to identify safe, tolerable, and clinically active dose (CAD) regimens of IMC-I109V for further clinical development. The IMC-I109V study is divided into 3 main parts: Part 1 - Single Ascending Dose (SAD); Part 2 - Multiple Ascending Dose (MAD), in HBeAg-negative CHB; Part 3 will evaluate safety, tolerability, antiviral activity, PK and anti-tumor efficacy of Multiple Ascending Doses of IMC-I109V in participants with HBV-associated hepatocellular carcinoma (HBV HCC) who are virally suppressed on NA therapy.

ELIGIBILITY:
Inclusion Criteria

Parts 1 and 2:

* ≥18 to 65 years old at time of informed consent
* HLA-A*02:01 positive
* Documented evidence of CHB based on one of the following: a. Positive HBsAg and HBV DNA at least 6 months prior to the Screening visit; OR b. Historical liver biopsy consistent with CHB infection.
* Have been receiving entecavir and/or tenofovir (including tenofovir alafenamide) for ≥12months prior to screening and are willing to continue.
* HBV DNA negative at screening
* No history of liver cirrhosis AND prior assessment of fibrosis demonstrating non-cirrhotic status at screening
* Participants of childbearing potential who are sexually active with a non-sterilized partner must agree to use highly effective methods of birth control from the trial screening date until 3 months after the final dose of the study intervention or longer if required by local regulations

Part 3:

* ≥18 years old at time of informed consent
* HLA-A*02:01 positive
* ECOG ≤1
* Locally advanced or metastatic and/or unresectable HCC with diagnosis confirmed by histology / cytology, or clinically by American Association for the Study of Liver Diseases criteria
* Failed or intolerant of ≥1 systemic therapy
* At least one measurable lesion (per RECIST 1.1) which is either not previously treated or, if treated, has clearly progressed prior to enrollment
* Documented evidence of CHB based on one of the following: a. Positive HBsAg and HBV DNA at least 6 months prior to the Screening visit; OR b. Historical liver biopsy consistent with CHB infection
* Life expectancy >3 months from time of enrolment
* Have compensated cirrhosis with a Child-Pugh score ≤ 7 (A or B7)
* On entecavir and/or tenofovir (disoproxil fumarate or alafenamide) with HBV DNA <100IU/ml at screening; willingness to continue for at least 6 months after the last dose of study drug
* Quantitative HBV surface antigen ≤ 5,000 IU/mL at screening
* Participants of childbearing potential who are sexually active with a non-sterilized partner must agree to use highly effective methods of birth control from the trial screening date until 3 months after the final dose of the study intervention or longer if required by local regulations

Exclusion Criteria:

Parts 1 and 2:

* Pregnant or lactating persons
* Known co-infection with any of the following: HIV, Hepatitis C virus, OR Hepatitis D virus
* Changes in HBeAg status within 3 months prior to the screening visit
* Known HBV genotype A
* Gilbert's syndrome
* Any known pre-existing medical or psychiatric condition that could interfere with the participant's ability to provide informed consent or participate in study conduct, or that may confound study findings including, but not limited to: Immunologically-mediated disease, e.g. inflammatory bowel disease (Crohn's disease, ulcerative colitis), rheumatoid arthritis, idiopathic thrombocytopenic purpura, systemic lupus erythematosus, scleroderma, or sarcoidosis within 5 years of the screening visit.
* Current or history of any clinically significant cardiac abnormalities/dysfunction, e.g. congestive heart failure, myocardial infarction ≤6 months prior to the screening visit, pulmonary hypertension, complex congenital heart disease, significant arrhythmia, or active cardiac ischemia.
* Evidence of decompensated liver disease including, but not limited to, a history or presence of clinical ascites, bleeding esophageal varices, hepatorenal syndrome, or hepatic encephalopathy.
* Significant immunosuppression from, but not limited to immunodeficiency conditions such as common variable hypogammaglobulinemia
* Evidence of active or suspected malignancy, or a history of malignancy ≤3 years prior to the screening visit (except adequately treated carcinoma in situ, basal cell carcinoma of the skin, or stage 0 HCC that has been treated). NOTE: Participants under evaluation for malignancy are not eligible
* Receiving or planning to receive systemic immunosuppressive medications during the study or ≤ 2 months prior to Day1, including but not limited to prednisone >10 mg/day (or equivalent), methotrexate, cyclosporine, or interferon. NOTE: Local steroid therapy is allowed (eg, inhaled, otic, ophthalmic, or intra-articular medications)
* Use of any live vaccines against infectious diseases within 4 weeks of the first planned administration of study intervention or use of any non-live vaccines against infectious diseases within 2 weeks of the first planned administration of study intervention.
* Treatment with any investigational drug or enrollment in any other clinical study ≤ 3 months prior to Day1, or at any time during participation in the study.
* Clinical diagnosis of substance abuse with alcohol, narcotics, or cocaine ≤12 months prior to the screening visit, except for those participants monitored in an opioid substitution maintenance program.

Part 3:

* Pregnant or lactating persons
* Untreated or symptomatic CNS metastases
* Significant ongoing toxicity from prior anticancer treatment -
* Ascites requiring recurrent paracentesis
* Inadequate washout from prior anticancer therapy
* Prior cellular therapy for HBV-associated HCC
* Known HBV genotype A
* Decompensated liver disease
* Surgical intervention or local / loco-regional therapy for HBV HCC within 28 days of planned first dose of study treatment
* Active hepatitis C virus (HCV) infection
* Untreated HIV infection
* Significant secondary malignancy
* Clinically significant lung, heart, or autoimmune disease
* Ongoing requirement for immunosuppressive treatment
* Prior solid organ or bone marrow transplant
* Hypersensitivity to study drug or excipients, or pre-medications
* Systemic antibiotics, vaccines or major surgery within 2-4 weeks prior to the first dose of study intervention
* Out-of-range laboratory values, including ALT or AST > 3x upper limit of normal (ULN), total bilirubin and direct bilirubin > 1.5x ULN, Albumin ≤ 28 g/L, International normalized ratio (INR) > 1.3

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2024-09-10 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Parts 1, 2, and 3: Incidence and treatment-emergent adverse events (TEAEs) | Up to 30 days after the last infusion of study treatment
Parts 1, 2, and 3: Incidence of serious adverse events (SAEs) | Up to 30 days after the last infusion of study treatment
Parts 1, 2, and 3: Incidence of adverse events (AEs) leading to treatment discontinuation | Up to 30 days after the last infusion of study treatment
Parts 1, 2, and 3: Incidence of dose-limiting toxicities (DLTs) | Up to 30 days after the last infusion of study treatment
Parts 1, 2, and 3: Changes in Vital Signs | Up to 30 days after the last infusion of study treatment
  Number of participants with, and rate of, Grade 1, Grade 2, Grade 3, and Grade 4 (as applicable per NCI CTCAE v5.0) vital sign abnormalities.
Parts 1, 2, and 3: Changes in electrocardiogram | Up to 30 days after the last infusion of study treatment
  QTcF interval absolute values and changes from baseline.
Parts 1, 2, and 3: Change in safety laboratory parameters | Up to 30 days after the last infusion of study treatment
  Number of participants with, and rate of, Grade 1, Grade 2, Grade 3, and Grade 4 (as applicable per NCI CTCAE v5.0) laboratory abnormalities.

SECONDARY OUTCOMES:
Parts 1, 2, and 3: Maximum drug concentration (Cmax) | At designated timepoints up to 162 days post-dose
Parts 1, 2, and 3: Area under the plasma concentration versus time curve (AUC) | At designated timepoints up to 162 days post-dose
Parts 1, 2, and 3: The time to reach maximum drug concentration (Tmax) | At designated timepoints up to 162 days post-dose
Parts 1, 2, and 3: The elimination half-life (t1/2) | At designated timepoints up to 162 days post-dose
Parts 1, 2, and 3: Incidence of anti-IMC-109V antibody formations | At designated timepoints up to 162 days post-dose
Parts 1, 2, and 3: Antiviral Effects: HBsAg change from baseline | Up to 280 days post-dose
Parts 1, 2, and 3: Antiviral Effects: HBcrAg change from baseline | Up to 280 days post-dose
Parts 1, 2, and 3: Antiviral Effects: HBV RNA change from baseline | Up to 280 days post-dose
Parts 1, 2, and 3: Antiviral Effects: HBsAb change from baseline | Up to 280 days post-dose
Part 3 only: Objective response rate (ORR) as determined by RECIST v1.1 as assessed by the Investigator | Up to ~52 months
Part 3 only: Overall survival (OS) as determined by RECIST v1.1 as assessed by the Investigator | Up to ~52 months
Part 3 only: Progression-free survival (PFS) as determined by RECIST v1.1 as assessed by the Investigator | Up to ~52 months
Part 3 only: Duration of response (DOR) as determined by RECIST v1.1 as assessed by the Investigator | Up to ~52 months

CONTACTS AND LOCATIONS:
Locations (15):
- United States (2):
  - University of Southern California Keck School of Medicine, Los Angeles, California
  - University Hospitals Cleveland Medical Center Case Western Reserve, Cleveland, Ohio
- Australia (2):
  - St. Vincent's Hospital, Fitzroy
  - The Alfred Centre, Melbourne
- Aarhus University, Aarhus, Denmark
- Queen Mary Hospital, Hong Kong, Hong Kong
- ARENSIA Exploratory Medicine Research Clinic, Bucharest, Romania
- Pusan National University Hospital, Busan, South Korea
- Spain (2):
  - Hospital Universitari Vall d'Hebron de Barcelona, Barcelona
  - Hospital Ramón and Cajal, Madrid
- Taiwan (2):
  - Kaohsiung Medical University Chung-Ho, Kaohsiung City
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (3):
  - Guy's Hospital, Dept. of Infectious Disease, London
  - Chelsea and Westminster Hospital, Research and Development, Clinical Trials Facility, London
  - Nottingham University Hospitals NHS Trust Biomedical Research Centre, Nottingham